CLINICAL TRIAL: NCT05269290
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled Study of the Efficacy and Safety of Ingavirin®, Syrup, 30 mg/5 ml, in Children Aged 6 Months to 2 Years With Influenza and Other Acute Respiratory Viral Infections Against Standard Therapy
Brief Title: Efficacy and Safety of Ingavirin®, Syrup, 30 mg/5 ml, in Children With Influenza and Other Acute Respiratory Viral Infections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Valenta Pharm JSC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ING-03-04-2020
Record Dates: First submitted 2022-01-28; First posted 2022-03-07 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Influenza, Human; Acute Respiratory Infection; Common Cold
MeSH Terms: conditions — Influenza, Human; Common Cold | interventions — pentanedioic acid imidazolyl ethanamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ingavirin®, syrup, 30 mg/5 ml (Experimental): Ingavirin®, syrup, 30 mg/5 ml will be administered on top of standard therapy
  Interventions: Drug: Ingavirin®, syrup, 30 mg/5 ml
- Placebo (Placebo Comparator): Placebo will be administered on top of standard therapy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ingavirin®, syrup, 30 mg/5 ml — A dose will be based on the body weight; Ingavirin® will be administered once a day on top of standard therapy.
  Arms: Ingavirin®, syrup, 30 mg/5 ml
Drug: Placebo — Placebo will be administered once a day on top of standard therapy.
  Arms: Placebo

SUMMARY:
The study is planned to evaluate the therapeutic efficacy and safety of Ingavirin®, syrup, 30 mg/5 ml, in the treatment of influenza or other acute respiratory infections in children from 6 months to 2 years compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Patient's parent/adoptive parent's informed consent form voluntarily signed by the patient's parent/adoptive parent;
2. Boys and girls aged 6 months - 2 years 11 months 14 days, inclusive, with the following clinical signs of acute respiratory infections/flu: body temperature above 38.0 °C but not higher than 39.0 °C (without taking antipyretics within the last 8 h) at the time of screening/randomization; at least one of the respiratory manifestations of acute respiratory infection/influenza (cough, runny nose/ stuffy nose) of at least 2 points on a 4-point scale; decrease in the child's daytime activity and change in nighttime sleep, as compared with the state before the illness;
3. There were no indications for hospitalization at the time of inclusion in the study;
4. Duration of illness from manifestation of symptoms to inclusion in the study not more than 48 hours.

Exclusion Criteria:

1. Presence of at least one of the epidemic signs: return from an overseas trip 14 days prior to the onset of symptoms; having close contact in the last 14 days with a person under observation for COVID-19 who has subsequently become ill; having close contact within the past 14 days with a person who has a laboratory-confirmed diagnosis of COVID-19;
2. Positive result of laboratory testing for SARS-CoV-2 RNA using nucleic acid amplification techniques or antigen SARS-CoV-2 antigen using an immunochromatographic assay at the time of screening;
3. Severe general intoxication syndrome (severe agitation with seizure syndrome and loss of consciousness against a background of hyperthermia);
4. Hemorrhagic syndrome (nasal bleeding, blood in sputum, vomit and stool, hemorrhagic rash), disseminated intravascular coagulation syndrome (DIC) or Hasser syndrome with the formation of acute renal failure;
5. Diffuse cyanosis or pallor;
6. Symptoms of pneumonia and possible acute respiratory distress syndrome (ARDS): cough with frothy sputum with blood, shortened pulmonary sound on percussion, a large number of different-caliber moist rales and abundant crepitation on auscultation, a sharp drop in blood pressure (BP), deafness of heart tones and arrhythmia;
7. Phenomena of respiratory distress combined with any of the following symptoms: grunting breathing, blowing of the wings of the nose when breathing, nodding movements (head movements synchronized with breathing); BPM in a child aged 6-11 months > 50 per minute, child over 1 year old > 40 per minute; lower chest retraction when breathing; blood oxygen saturation (SpO2) < 92% when breathing room air;
8. Moderate acute respiratory infections (fever ≥ 38.5 °C) with exacerbation of comorbidities;
9. Presence of any of the following symptoms: inability to drink/breastfeed; drowsiness or unconsciousness; respiratory rate less than 30 per minute or apnea; heart failure phenomena; severe dehydration;
10. Febrile seizures, including a history of seizures; known intolerance to the active ingredient or excipient of the study drug or placebo components, paracetamol;

12. Lactose intolerance, lactase deficiency or glucose-galactose malabsorption. 13. Taking antibiotics, antivirals, or immunomodulatory drugs within < 48 h prior to the study and/or plans to use these groups of drugs (other than the study drug) during the study; 14. Use of systemic, inhaled, or nasal glucocorticosteroids within 30 days prior to the study and/or plans to use glucocorticosteroids (except topical cutaneous agents) during the study; 15. Failure to withdraw for the duration of the study other medications that may affect the outcome of this study, such as antiviral medications, or medications that are incompatible with the study therapy (see "prohibited concomitant therapies"); 16. Patient's participation in any other clinical trial within 90 days prior to inclusion in the study; 17. Any cardiovascular, renal, hepatic, gastrointestinal (GI), endocrine, or nervous system disease, severe decompensated chronic or acute disease, or any other condition/disease that, in the opinion of the investigating physician, would make it unsafe for the patient to participate in the study; 18. Having any vaccinations administered to the patient within 14 days prior to inclusion in the study; 19. Diabetes mellitus; 20. Clinical suspicion of pneumonia or other bacterial infections (including sinusitis, otitis media, urinary tract infection, meningitis, sepsis, etc.) requiring administration of antibacterial drugs; 21. Patients who have had surgery within 30 days prior to the Screening Visit and patients who are scheduled to have surgery, including diagnostic procedures, or a hospital stay during the study; 22. Suspicion of hemophagocytic syndrome; 23. Increased seizure activity in the history; 24. The presence of cancer, HIV infection, tuberculosis, including in the anamnesis; 25. Suspected low compliance of the parent/adopter with the child's treatment and recording of required parameters in the Patient Diary, or inability to perform these procedures and comply with restrictions according to the study protocol (e.g., due to mental illness).

Withdrawal Criteria:

1. Identification of a probable or confirmed case COVID-19;
2. Signs of complications of viral infection, including signs of secondary bacterial infection;
3. The investigating physician decides that the patient must be excluded for the patient's own benefit;
4. Withdrawal of informed consent by the parent or adoptive parent;
5. Individual intolerance to the study drug;
6. Development of NS requiring withdrawal of study drug/placebo;
7. Erroneous inclusion (for example, the patient was included in violation of the inclusion/inclusion criteria of the protocol);
8. Patient receives/needs additional treatment that may affect study outcome or patient safety (see "prohibited concomitant therapies");
9. Persistence of nasal congestion longer than 10 days, worsening of condition after the first week of illness, facial pain;
10. Patient's development of the conditions described in the criteria for exclusion;
11. Development of hemorrhagic syndrome (including DIC): nosebleed, hemorrhagic rash on the face, neck, chest, and upper extremities, hemorrhages into the mucous membrane of the mouth and nose, the back of the throat, conjunctivae, blood in vomit, hemoptysis, etc.);
12. A pronounced intoxication syndrome with the development of encephalic or meningoencephalic reactions (delirium, hallucinations, seizures, confusion or loss of consciousness, vomiting);
13. Hemophagocytic syndrome;
14. Other conditions or events that, in the opinion of the investigating physician, require exclusion of the patient from the study.

Ages: 6 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Time of symptoms/events resolution | From Day 1 up to Day 13-14 (visit 4)
  Time, in hours, from the first administration of the drug until all of the following symptoms/events have resolved (if each symptom/event has been achieved for at least 24 hours): Fever; Cough and/or runny nose/nasal congestion; Child's return to normal daytime activity and normal nighttime sleep (as assessed by the parent/adopter).

SECONDARY OUTCOMES:
Time to fever relief | From Day 1 up to Day 13-14 (visit 4)
  Number of hours elapsed from the first administration of the medication to the time of persistent normalization of the temperature, i.e., the moment when the body temperature is < 37.5 °C during the day without the use of antipyretic medication
Time to cough relief | From Day 1 up to Day 13-14 (visit 4)
  Number of hours from the first dose to the time the coughing cough has gone away, i.e. the parent/adoptive parent rates the symptom as 0-1 during the day and records this in the patient's diary
Time to cough/nasal congestion relief | From Day 1 up to Day 13-14 (visit 4)
  Number of hours from first medication administration to cough/congestion cessation, i.e., when parent/adopter rates severity of this symptom during the day at 0-1 point and records this in patient diary
Frequency of complications of acute viral infection and influenza | From Day 1 up to Day 13-14 (visit 4)
  Acute otitis media, viral and bacterial pneumonia, exacerbation of chronic conditions such as bronchial asthma and urinary tract infections), toxemia [septic-like syndrome], acute stenotic laryngotracheitis
Frequency of patients with PCR-confirmed viral infection | Day 1, Day 3-4 (visit 2), Day 6-7 (visit 3)
  PCR-confirmed acute respiratory infections/flu by visits 1, 2, 3
Need for paracetamol or ibuprofen | Days 1-7
  Daily dose on study days 1-7
Safety - Number of adverse events (AEs) | From Day 1 up to Day 13-14 (visit 4) or up to early termination visit within time frame of the study
  Total number of AEs stratified by severity and frequency
Safety - Adverse reactions | From Day 1 up to Day 13-14 (visit 4) or up to early termination visit within time frame of the study
  Frequency of adverse reactions
Safety - Serious adverse events (SAEs) | From Day 1 up to Day 13-14 (visit 4) or up to early termination visit within time frame of the study
  Frequency of serious adverse events (SAEs) associated with study drug/placebo use
Safety - Percentage of patients with AEs | From Day 1 up to Day 13-14 (visit 4) or up to early termination visit within time frame of the study
  Percentage of patients with at least one AE
Safety - Percentage of patients who interrupted treatment | From Day 1 up to Day 13-14 (visit 4) or up to early termination visit within time frame of the study
  Percentage of patients who interrupted treatment due to AE
Safety - Frequency of complications | From Day 1 up to Day 13-14 (visit 4) or up to early termination visit within time frame of the study
  Frequency of complications
Safety - Frequency of worsening | From Day 1 up to Day 13-14 (visit 4) or up to early termination visit within time frame of the study
  Frequency of worsening of the disease course
Safety - Frequency of hospitalization | From Day 1 up to Day 13-14 (visit 4) or up to early termination visit within time frame of the study
  Frequency of need for hospitalization

CONTACTS AND LOCATIONS:
Locations (8):
- Russia (8):
  - Federal Research and Clinical Center of Physical and Chemical Medicine of the Federal Medical and Biological Agency, Odintsovo, Moscow Oblast
  - City Pediatric Outpatient Clinic number 5, Perm
  - Professors' Clinic LLC., Perm
  - St. Petersburg State Budgetary Healthcare Institution "Children's City Polyclinic No. 44", Saint Petersburg
  - City Polyclinic No. 45 of Nevsky District, Saint Petersburg
  - PiterKlinika LLC, Saint Petersburg
  - Uromed LLC, Smolensk
  - Bashkir State Medical University, Ufa

IPD SHARING:
Plan to Share IPD: Undecided